CLINICAL TRIAL: NCT03164460
Title: Phase II Randomized Trial of Stereotactic Onco-Ablative Reirradiation Versus Conventionally Fractionated Conformal Radiotherapy for Patients With Small Inoperable Head and Neck Tumors (SOAR-HN)
Brief Title: Stereotactic Body Radiation Therapy or Intensity Modulated Radiation/Proton Therapy in Treating Patients With Recurrent Head and Neck Cancer
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: DMC Monitor Action
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1065; NCI-2018-01190 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-1065 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Head and Neck Carcinoma
MeSH Terms: interventions — Radiotherapy, Intensity-Modulated; Proton Therapy; Radiation; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (SBRT) (Experimental): Patients undergo SBRT every other day for a total of 5 treatments.
  Interventions: Radiation: Stereotactic Body Radiation Therapy
- Group II (IMRT/IMPT) (Experimental): Patients undergo IMRT/IMPT once daily (Monday-Friday) for up to 30-35 treatments.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy; Radiation: Proton Radiation

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT/IMPT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
  Arms: Group II (IMRT/IMPT)
Radiation: Proton Radiation — Undergo IMRT/IMPT
  Other Names: Radiation, Charged Particles-Protons
  Arms: Group II (IMRT/IMPT)
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Group I (SBRT)

SUMMARY:
This phase II trial studies how well stereotactic body radiation therapy or intensity modulated radiation/proton therapy works in treating patients with head and neck cancer that has come back. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Intensity modulated radiation/proton therapy uses high energy x-rays or protons to kill tumor cells and shrink tumors. It is not yet known whether stereotactic body radiation therapy or intensity modulated radiation/proton therapy may work better in treating patients with head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the 2-year rate of Common Terminology Criteria for Adverse Events (CTCAE)-4.0 grade 3 or higher toxicity at 2 years between the two treatment arms.

SECONDARY OBJECTIVES:

I. To compare the 2-year locoregional failure free survival (LFFS) in patients being treated with reirradiation with either stereotactic ablative radiotherapy (SBRT) versus intensity modulated radiation therapy/intensity modulated proton therapy (IMRT/IMPT).

II. To determine if there is any difference in local control, progression-free survival, and overall survival between the two arms.

III. To compare toxicity using Common Terminology Criteria for Adverse Events (CTCAE)-4.0 and Performance Status Scale-HN (Head and Neck).

IV. To compare patient reported outcome (PRO) measures of symptoms using MD Anderson Symptom Inventory (MDASI), MD Anderson Dysphagia Inventory (MDADI), Functional Assessment of Cancer Therapy (FACT)-HN, ACT-HN Symptom Index (FACT-HNSI), MD Anderson Symptom Inventory-Brain Tumor (MDASI-BT), for skull base only, Anterior Skull BASE Questionnaire (ASBQ), for skull base only, Brief Fatigue Inventory (BFI), Telephone Interview for Cognitive Status (TICS), Performance Status Scale For Head and Neck Cancer Patients (PSS-HN), Work Productivity and Activity Impairment Questionnaire: Specific Health Problem version (V)2.0 (WPAI:SHP), and University of Michigan Xerostomia-Related Quality of Life Scale, Xerostomia and Health Questionnaire (European Quality of Life Five Dimension Three Level [EQ-5D-3L]).

V. Quality-Adjusted-Life-Years (QALY) comparison between IMPT and IMRT. VI. Compare cost-benefit economic analysis of treatment. VII. Perform dosimetric analysis and compare correlates of critical structures.

EXPLORATORY OBJECTIVES:

I. To assess potential differences between patients on study and patients who were considered eligible for randomized, were randomized to a treatment arm, but may have dropped out of the study for other reasons after being randomized to; or were denied insurance coverage for the treatment arm she/he was randomized.

OUTLINE: Patients are randomized into 1 of 2 groups.

GROUP I: Patients undergo SBRT every other day for a total of 5 treatments.

GROUP II: Patients undergo IMRT/IMPT once daily (Monday-Friday) for up to 30-35 treatments.

After completion of study treatment, patients are followed up at 2-3 months, every 3 months for 1 year, and then every 3-4 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented recurrent head and neck cancer, or second primary head and neck cancer, AND who have previously received radiation (at least 30 Gy) for head and neck cancer
* Not eligible for surgery for recurrence or poor surgical candidate
* Gross disease apparent on imaging (magnetic resonance imaging [MRI] or computed tomography [CT])
* 1-3 sites of recurrence (< 60 cc per site, total volume < 100 cc)
* Eastern Cooperative Oncology Group (ECOG) = 0, 1, or 2
* Negative pregnancy test for women of child bearing potential

Exclusion Criteria:

* Patients who are pregnant or breast feeding
* Clinically significant uncontrolled major cardiac, respiratory, renal, hepatic, gastrointestinal or hematologic disease but not limited to:

  * a) Symptomatic congestive heart failure, unstable angina, or cardiac dysrhythmia not controlled by pacer device
  * b) No myocardial infarction within 3 months of registration
* Widely metastatic disease (oligometastatic disease acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3+ toxicity (Tox3+) assessed by Common Terminology Criteria for Adverse Events (CTCAE) | At 2 years
  Will use the methods of Gooley et al. to estimate the cumulative incidence of Tox3+, as well as competing-risk regression to model cumulative incidence of Tox3+ while treating death not related to Tox3+ as a competing event. The student t-test or the Wilcoxon rank sum test will be used to compare continuous variables between patient groups. The chi-square test or the Fisher's exact test will be applied to evaluate the association between two categorical variables. Logistic regression models will be used to evaluate the effects of the important patient clinical factors including treatment on TOX3+.

SECONDARY OUTCOMES:
Local control defined as absence of local failure | Up to 2 years
  The student t-test or the Wilcoxon rank sum test will be used to compare continuous variables between patient groups. The chi-square test or the Fisher's exact test will be applied to evaluate the association between two categorical variables. Logistic regression models will be used to evaluate the effects of the important patient clinical factors including treatment on TOX3+.
Local failure free survival (LFFS) defined as failure (recurrence or progression) within the prescribed radiation field, including failure within 2 cm of the radiation field | From treatment initiation until local failure or death from any cause, assessed at 2 years
  Will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test. Proportional hazards regression may be employed for multivariate analysis on time-to-event outcomes.
Incidence of acute grade 3 or higher toxicity assessed by CTCAE | Up to 90 days after completion of radiation therapy
  The student t-test or the Wilcoxon rank sum test will be used to compare continuous variables between patient groups. The chi-square test or the Fisher's exact test will be applied to evaluate the association between two categorical variables. Logistic regression models will be used to evaluate the effects of the important patient clinical factors including treatment on TOX3+.
Incidence of late grade 3 or higher toxicity assessed by CTCAE | 90 days up to 2 years
  The student t-test or the Wilcoxon rank sum test will be used to compare continuous variables between patient groups. The chi-square test or the Fisher's exact test will be applied to evaluate the association between two categorical variables. Logistic regression models will be used to evaluate the effects of the important patient clinical factors including treatment on TOX3+.
Progression free survival (PFS) | From treatment initiation until an LFFS event, or occurrence, recurrence, or progression of distant metastases, whichever occurs first, assessed up to 2 years
  PFS event is defined as an LFFS event, or occurrence, recurrence or progression of distant metastases. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test. Proportional hazards regression may be employed for multivariate analysis on time-to-event outcomes.
Overall survival | From treatment initiation until time to death from any cause, assessed up to 2 years
  Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test. Proportional hazards regression may be employed for multivariate analysis on time-to-event outcomes.
Patient reported outcomes (PROs) | Up to 2 years
  Generalized linear models for the repeated measures analysis will be performed to assess the change in PROs overtime with important covariates including treatment in the models.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Phan, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org